CLINICAL TRIAL: NCT04234854
Title: OPTIMAl Endovascular Exclusion of High-risk Carotid Plaque Using the CGuard™ Stent in Patients With Symptoms or Signs of Carotid Stenosis-related Brain Injury: IVUS Controlled Investigator Initiated Multcentric Multi-specialty Study
Brief Title: OPTIMAl Endovascular Exclusion of Consecutive Patient High-risk Carotid Plaque Using the MicroNet Covered Stent
Acronym: OPTIMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: John Paul II Hospital, Krakow (Other)
Collaborators: InspireMD (Industry)
Responsible Party: Sponsor
Other Study IDs: OPTIMA
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Carotid Artery Diseases
Keywords: Stenting
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carotid Artery Stenting: Consecutive patients older than 18 yrs with symptomatic carotid artery stenosis qualified for endovascular revascularization.
  Interventions: Diagnostic Test: Intravascular Utrasound (IVUS) of Carotid Artery after implantation of CGuard stent

INTERVENTIONS:
Diagnostic Test: Intravascular Utrasound (IVUS) of Carotid Artery after implantation of CGuard stent — IVUS will be performed after stent postdilatation to determine the incidence of plaque prolapse. Additionally optimizing stent expansion with IVUS is left at operator discretion.

SUMMARY:
Prospective, multicentric, multispecialty, international, open-label, single arm study using per-protocol intravascular ultrasound [IVUS, 20MHz electronic phase-array transducer] to document the procedure result of an effective plaque exclusion from the vessel lumen.

DETAILED DESCRIPTION:
Investigator initiated, academic, single arm, open-label, non-randomized, prospective, multicenter, multispecialty trial of CGuard™ use in all-comer population of consecutive patients with carotid stenosis related cerebral symptoms (TIA, stroke, retinal TIA, retinal stroke) or signs of ipsilateral brain injury on MRI or CT imaging.

The main objective of this observational study is to evaluate an incidence of residual plaque prolapse after carotid stenting using the study device.

Study Rationale In conventional carotid stents, plaque prolapse (PP) on intravascular imaging had been determined to be strongly associated with new post-procedural diffusion-weighted magnetic resonance lesions on cerebral imaging and with increased ischaemic stroke incidence. A significant increase in PP susceptibility was observed with unstable carotid plaque, pointing to the limitations of conventional CAS in unstable carotid plaques, such as symptomatic and increased-spontaneous-symptoms-risk lesions.

This is reflected in current guidelines that provide a higher recommendation class to surgical management (CEA) rather than CAS for symptomatic lesions.

Circumstantial evidence indicates that the novel carotid stent covered with MicroNET (CGuard EPS) may be an optimal device for effective carotid plaque sequestration (that may be particularly relevant in high-risk plaques) - but no systematic study has been performed thus far.

Because of the increasing evidence that not only clinical symptoms (that may be related to for instance the affection of dominant vs. non-dominant haemisphere) but also signs of ipisilateral cerebral infarct/s are a hallmark of high-risk plaque and are associated with adverse prognosis, and because that neurology increasingly uses the term "symptomatic" to refer to carotid stenosis associated with clinically silent ipisilateral cerebral infarct/s, the present study will enroll both patients with clinical symptoms of cerebral ischaemia in relation to carotid stenosis and those with (clinically silent) signs of ipsilateral injury such as ischemic focus/foci on CT or MRI/DW-MRI).

As previously demonstrated, clinically significant/relevant PP is that depicted by IVUS (with angiography, on the one hand, being not sensitive enough and OCT, on the other, being possibly too sensitive).

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients with clinically symptomatic carotid stenosis , or carotid stenosis associated with ipisilateral cerebral ischemic infarct/s on CT or MRI/DWI imaging, referred and accepted by the study center for CAS as per local standard referral pathways and study center routine.
* Patient informed consent to participate.
* Patient accepts follow-up scheme and consents to follow-up visits.

Exclusion Criteria:

* Lack of indication to carotid revascularization as per current ESC/ESVS Guidelines, or any clinical or angiographic or other contraindication to CAS (such as renal failure defined as creatinine level > 2.5 mg/dL or eGFR <20 ml/kg min, or incompatibility with DAPT).
* Surgery within the preceding 30 days or planned surgery within 30 days after CAS.
* Life expectancy <1 year (eg. neoplastic disease).
* MI within 72h prior to CAS.
* Known coagulopathy.
* History of cerebral stroke with documented/known cause other than carotid disease.
* Atrial fibrillation or flutter.
* Any known cause for potential cerebral embolization different than carotid stenosis.
* History of intracranial bleeding.
* Any contraindications to as per IFU study device implantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive clinically-symptomatic patients (ipsilateral cerebral or retinal stroke or TIA with the preceding 6 months) with atherosclerotic de novo carotid artery stenosis causing at least 50% lumen reduction by quantitative carotid catheter angiography (QCA) or carotid stenosis of at least 50% lumen reduction by QCA in relation to documented ipsilateral ischaemic brain lesions/infarct on CT or MRI.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Freedom from plaque prolapse | During index procedure
  Freedom from plaque prolapse defined as observation of plaque inside the stent lumen after completion of the CAS procedure by IVUS assessment (Kotsugi 2017).

SECONDARY OUTCOMES:
Procedural success | During index procedure
  stent delivery and implantation in absence of an intra-procedural clinical major adverse event, with no more than 30% residual diameter stenosis by on-site QCA, and successful withdrawal of the stent delivery and neuroprotection system
IVUS interrogation success | During index procedure
  IVUS interrogation with an effective IVUS probe removal in absence of any clinical complications
Endovascular lumen reconstruction | During index procedure
  Freedom from plaque prolapse plus minimal in-stent area >50% ICA reference area
Periprocedural MACCE | Until discharge or up to 24 hours
  Death, stroke, myocardial infarction until discharge or up to 24 hours
30 days MACCE | 30 days
  Death, stroke, myocardial infarction until 30 days
Any periprocedural complications | Until discharge or up to 24 hours
  Any complications occurring until discharge or 24 hours whichever comes first
Ipsilateral stroke between 31 days and 12 months after the procedure | Between 31 days and 12 months after the procedure
  Ipsilateral stroke between 31 days and 12 months after the procedure
Duplex UltraSound (DUS) at 30 days | 30 days
  Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV) recorded by Duplex Doppler at 30±5 days after the procedure
Duplex UltraSound (DUS) at 12 months | 12 months
  Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV) recorded by Duplex Doppler at 12 months after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Musialek, MD, PhD, Study Chair — Department of Cardiac and Vascular Diseases, The John Paul II Hospital
Locations (1):
- Department of Cardiac and Vascular Diseases, The John Paul II Hospital, Krakow, Maloplska, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kotsugi M, Takayama K, Myouchin K, Wada T, Nakagawa I, Nakagawa H, Taoka T, Kurokawa S, Nakase H, Kichikawa K. Carotid Artery Stenting: Investigation of Plaque Protrusion Incidence and Prognosis. JACC Cardiovasc Interv. 2017 Apr 24;10(8):824-831. doi: 10.1016/j.jcin.2017.01.029. PMID 28427600
- [Background] Musialek P, Pieniazek P, Tracz W, Tekieli L, Przewlocki T, Kablak-Ziembicka A, Motyl R, Moczulski Z, Stepniewski J, Trystula M, Zajdel W, Roslawiecka A, Zmudka K, Podolec P. Safety of embolic protection device-assisted and unprotected intravascular ultrasound in evaluating carotid artery atherosclerotic lesions. Med Sci Monit. 2012 Feb;18(2):MT7-18. doi: 10.12659/msm.882452. PMID 22293887
- [Background] Clark DJ, Lessio S, O'Donoghue M, Schainfeld R, Rosenfield K. Safety and utility of intravascular ultrasound-guided carotid artery stenting. Catheter Cardiovasc Interv. 2004 Nov;63(3):355-62. doi: 10.1002/ccd.20188. PMID 15505835
- [Background] Bandyk DF, Armstrong PA. Use of intravascular ultrasound as a "Quality Control" technique during carotid stent-angioplasty: are there risks to its use? J Cardiovasc Surg (Torino). 2009 Dec;50(6):727-33. PMID 19935603
- [Background] Hitchner E, Zhou W. Utilization of Intravascular Ultrasound during Carotid Artery Stenting. Int J Angiol. 2015 Sep;24(3):185-8. doi: 10.1055/s-0035-1556081. Epub 2015 Jul 10. PMID 26417186
- [Background] Musialek P, Hopf-Jensen S. Commentary: Carotid Artery Revascularization for Stroke Prevention: A New Era. J Endovasc Ther. 2017 Feb;24(1):138-148. doi: 10.1177/1526602816671263. Epub 2016 Oct 13. No abstract available. PMID 27733691
- [Background] Schofer J, Musialek P, Bijuklic K, Kolvenbach R, Trystula M, Siudak Z, Sievert H. A Prospective, Multicenter Study of a Novel Mesh-Covered Carotid Stent: The CGuard CARENET Trial (Carotid Embolic Protection Using MicroNet). JACC Cardiovasc Interv. 2015 Aug 17;8(9):1229-1234. doi: 10.1016/j.jcin.2015.04.016. PMID 26292586
- [Background] Musialek P, Mazurek A, Trystula M, Borratynska A, Lesniak-Sobelga A, Urbanczyk M, Banys RP, Brzychczy A, Zajdel W, Partyka L, Zmudka K, Podolec P. Novel PARADIGM in carotid revascularisation: Prospective evaluation of All-comer peRcutaneous cArotiD revascularisation in symptomatic and Increased-risk asymptomatic carotid artery stenosis using CGuard MicroNet-covered embolic prevention stent system. EuroIntervention. 2016 Aug 5;12(5):e658-70. doi: 10.4244/EIJY16M05_02. PMID 27180302
- [Background] Ruffino MA, Faletti R, Fronda M, Gatti M, Bergamasco L, Gibello L, Varetto G, Righi D, Rispoli P, Fonio P. Early Embolization After Carotid Artery Stenting with Mesh-Covered Stent: Role of Diffusion-Weighted Magnetic Resonance Imaging as Pre-procedural Predictor and Discriminant Between Intra- and Post-procedural Events. Cardiovasc Intervent Radiol. 2019 Jun;42(6):812-819. doi: 10.1007/s00270-019-02173-1. Epub 2019 Feb 19. PMID 30783778
- [Background] Speziale F, Capoccia L, Sirignano P, Mansour W, Pranteda C, Casana R, Setacci C, Accrocca F, Alberti D, de Donato G, Ferri M, Gaggiano A, Galzerano G, Ippoliti A, Mangialardi N, Pratesi G, Ronchey S, Ruffino A, Siani A, Spinazzola A, Sponza M. Thirty-day results from prospective multi-specialty evaluation of carotid artery stenting using the CGuard MicroNet-covered Embolic Prevention System in real-world multicentre clinical practice: the IRON-Guard study. EuroIntervention. 2018 Feb 20;13(14):1714-1720. doi: 10.4244/EIJ-D-17-00008. PMID 28485278
- [Background] Musialek P, Grunwald IQ. How asymptomatic is "asymptomatic" carotid stenosis? Resolving fundamental confusion(s) - and confusions yet to be resolved. Pol Arch Intern Med. 2017 Nov 30;127(11):718-719. doi: 10.20452/pamw.4157. Epub 2017 Nov 30. No abstract available. PMID 29192895
- [Background] Stabile E, Sannino A, Schiattarella GG, Gargiulo G, Toscano E, Brevetti L, Scudiero F, Giugliano G, Perrino C, Trimarco B, Esposito G. Cerebral embolic lesions detected with diffusion-weighted magnetic resonance imaging following carotid artery stenting: a meta-analysis of 8 studies comparing filter cerebral protection and proximal balloon occlusion. JACC Cardiovasc Interv. 2014 Oct;7(10):1177-83. doi: 10.1016/j.jcin.2014.05.019. Epub 2014 Sep 17. PMID 25240544
- [Background] Wissgott C, Schmidt W, Brandt-Wunderlich C, Behrens P, Andresen R. Clinical Results and Mechanical Properties of the Carotid CGUARD Double-Layered Embolic Prevention Stent. J Endovasc Ther. 2017 Feb;24(1):130-137. doi: 10.1177/1526602816671134. Epub 2016 Oct 13. PMID 27733689
- [Background] Stabile E, de Donato G, Musialek P, De Loose K, Nerla R, Sirignano P, Chianese S, Mazurek A, Tesorio T, Bosiers M, Setacci C, Speziale F, Micari A, Esposito G. Use of Dual-Layered Stents in Endovascular Treatment of Extracranial Stenosis of the Internal Carotid Artery: Results of a Patient-Based Meta-Analysis of 4 Clinical Studies. JACC Cardiovasc Interv. 2018 Dec 10;11(23):2405-2411. doi: 10.1016/j.jcin.2018.06.047. PMID 30522670
- [Background] Casana R, Tolva V, Odero A Jr, Malloggi C, Paolucci A, Triulzi F, Silani V. Safety and Efficacy of the New Micromesh-Covered Stent CGuard in Patients Undergoing Carotid Artery Stenting: Early Experience From a Single Centre. Eur J Vasc Endovasc Surg. 2017 Dec;54(6):681-687. doi: 10.1016/j.ejvs.2017.09.015. Epub 2017 Oct 28. PMID 29089282
- [Background] Umemoto T, de Donato G, Pacchioni A, Reimers B, Ferrante G, Isobe M, Setacci C. Optical coherence tomography assessment of newgeneration mesh-covered stents after carotid stenting. EuroIntervention. 2017 Dec 20;13(11):1347-1354. doi: 10.4244/EIJ-D-16-00866. PMID 28760722
- [Background] de Donato G, Setacci F, Sirignano P, Galzerano G, Cappelli A, Setacci C. Optical coherence tomography after carotid stenting: rate of stent malapposition, plaque prolapse and fibrous cap rupture according to stent design. Eur J Vasc Endovasc Surg. 2013 Jun;45(6):579-87. doi: 10.1016/j.ejvs.2013.03.005. Epub 2013 Apr 10. PMID 23582886
- [Background] Umemoto T, Pacchioni A, Nikas D, Reimers B. Recent developments of imaging modalities of carotid artery stenting. J Cardiovasc Surg (Torino). 2017 Feb;58(1):25-34. doi: 10.23736/S0021-9509.16.09813-X. Epub 2016 Dec 6. PMID 27922253
- [Background] de Donato G, Setacci C, Umemoto T, Reimers B. Commentary: Inside of the Interaction Between the Plaque and the Stent: Optical Coherence Tomography During Carotid Artery Stenting. J Endovasc Ther. 2015 Dec;22(6):950-1. doi: 10.1177/1526602815611885. No abstract available. PMID 26586654
- [Background] Musialek P, Stabile E. Residual plaque prolapse with novel dual-layer carotid stents: is it mesh-covered or not? EuroIntervention. 2017 Dec 20;13(11):1266-1268. doi: 10.4244/EIJV13I11A199. No abstract available. PMID 29260718
- [Background] Pacchioni A, Ribichini F, Reimers B. Stent Type and Risk of Late Cerebral Events After Carotid Artery Stenting. J Am Coll Cardiol. 2015 Jul 28;66(4):490. doi: 10.1016/j.jacc.2015.04.074. No abstract available. PMID 26205606
- [Background] Secco GG, Cremonesi A, Amor M, Pistis G, Reimers B, Castriota F. Optical coherence tomography during carotid artery stenting: A new niche application? Int J Cardiol. 2015;187:372-3. doi: 10.1016/j.ijcard.2015.03.237. Epub 2015 Mar 18. No abstract available. PMID 25841129
- [Background] Musialek P, Hopkins LN, Siddiqui AH. One swallow does not a summer make but many swallows do: accumulating clinical evidence for nearly-eliminated peri-procedural and 30-day complications with mesh-covered stents transforms the carotid revascularisation field. Postepy Kardiol Interwencyjnej. 2017;13(2):95-106. doi: 10.5114/pwki.2017.69012. Epub 2017 Jul 19. PMID 28798779
- [Background] Aboyans V, Ricco JB, Bartelink MEL, Bjorck M, Brodmann M, Cohnert T, Collet JP, Czerny M, De Carlo M, Debus S, Espinola-Klein C, Kahan T, Kownator S, Mazzolai L, Naylor AR, Roffi M, Rother J, Sprynger M, Tendera M, Tepe G, Venermo M, Vlachopoulos C, Desormais I, Document Reviewers, Widimsky P, Kolh P, Agewall S, Bueno H, Coca A, De Borst GJ, Delgado V, Dick F, Erol C, Ferrini M, Kakkos S, Katus HA, Knuuti J, Lindholt J, Mattle H, Pieniazek P, Piepoli MF, Scheinert D, Sievert H, Simpson I, Sulzenko J, Tamargo J, Tokgozoglu L, Torbicki A, Tsakountakis N, Tunon J, Vega de Ceniga M, Windecker S, Zamorano JL. Editor's Choice - 2017 ESC Guidelines on the Diagnosis and Treatment of Peripheral Arterial Diseases, in collaboration with the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2018 Mar;55(3):305-368. doi: 10.1016/j.ejvs.2017.07.018. Epub 2017 Aug 26. No abstract available. PMID 28851596
- [Background] Naylor AR, Ricco JB, de Borst GJ, Debus S, de Haro J, Halliday A, Hamilton G, Kakisis J, Kakkos S, Lepidi S, Markus HS, McCabe DJ, Roy J, Sillesen H, van den Berg JC, Vermassen F, Esvs Guidelines Committee, Kolh P, Chakfe N, Hinchliffe RJ, Koncar I, Lindholt JS, Vega de Ceniga M, Verzini F, Esvs Guideline Reviewers, Archie J, Bellmunt S, Chaudhuri A, Koelemay M, Lindahl AK, Padberg F, Venermo M. Editor's Choice - Management of Atherosclerotic Carotid and Vertebral Artery Disease: 2017 Clinical Practice Guidelines of the European Society for Vascular Surgery (ESVS). Eur J Vasc Endovasc Surg. 2018 Jan;55(1):3-81. doi: 10.1016/j.ejvs.2017.06.021. Epub 2017 Aug 26. No abstract available. PMID 28851594
- [Background] Morr S, Vakharia K, Fanous AA, Waqas M, Siddiqui AH. Utility of Intravascular Ultrasound During Carotid Angioplasty and Stenting with Proximal Protection. Cureus. 2019 Jun 18;11(6):e4935. doi: 10.7759/cureus.4935. PMID 31431840
- [Background] Chiocchi M, Morosetti D, Chiaravalloti A, Loreni G, Gandini R, Simonetti G. Intravascular ultrasound assisted carotid artery stenting: randomized controlled trial. Preliminary results on 60 patients. J Cardiovasc Med (Hagerstown). 2019 Apr;20(4):248-252. doi: 10.2459/JCM.0b013e32835898f1. PMID 23292649
- [Background] Joan MM, Moya BG, Agusti FP, Vidal RG, Arjona YA, Alija MP, Paredero VM. Utility of intravascular ultrasound examination during carotid stenting. Ann Vasc Surg. 2009 Sep-Oct;23(5):606-11. doi: 10.1016/j.avsg.2008.09.010. Epub 2009 Jun 24. PMID 19556101
- [Background] Wehman JC, Holmes DR Jr, Ecker RD, Sauvageau E, Fahrbach J, Hanel RA, Hopkins LN. Intravascular ultrasound identification of intraluminal embolic plaque material during carotid angioplasty with stenting. Catheter Cardiovasc Interv. 2006 Dec;68(6):853-7. doi: 10.1002/ccd.20871. PMID 17086527
- [Background] Musialek P, Roubin GS. Commentary: Double-Layer Carotid Stents: From the Clinical Need, through a Stent-in-Stent Strategy, to Effective Plaque Isolation... the Journey Toward Safe Carotid Revascularization Using the Endovascular Route. J Endovasc Ther. 2019 Aug;26(4):572-577. doi: 10.1177/1526602819861546. No abstract available. PMID 31303133